CLINICAL TRIAL: NCT05665751
Title: A Phase 2a Study Evaluating the Safety, Tolerability, and Efficacy of TLC-3595 in Subjects With Insulin Resistance
Brief Title: A Study Evaluating Daily Oral Doses of TLC-3595 in Participants With Insulin Resistance
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: OrsoBio, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3595-CL-101
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TLC-3595 Dose 1 (Experimental): Oral dose of TLC-3595 Dose 1
  Interventions: Drug: TLC-3595 Dose 1
- TLC-3595 Dose 2 (Experimental): Oral dose of TLC-3595 Dose 2
  Interventions: Drug: TLC-3595 Dose 2
- Placebo (Placebo Comparator): Oral dose of placebo-to-match
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TLC-3595 Dose 1 — Tablets administered orally
  Arms: TLC-3595 Dose 1
Drug: TLC-3595 Dose 2 — Tablets administered orally
  Arms: TLC-3595 Dose 2
Drug: Placebo — Tablets administered orally
  Arms: Placebo

SUMMARY:
This Phase 2a study is designed to evaluate the safety, tolerability, effectiveness, and pharmacokinetics (PK) of TLC-3595 in subjects with insulin resistance.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized study. Participants will be randomized to one of three treatment arms, to receive one of the two doses of TLC-3595 (or matching placebo).

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 18-70 years of age, inclusive, at Screening
* BMI ≥ 28 kg/m2 at Screening
* Diagnosis of insulin resistance based on HOMA-IR > 2.84 at Screening or a confirmed diagnosis of type 2 diabetes mellitus
* Screening laboratory evaluations (hematology, chemistry, and urinalysis) must fall within the protocol-defined ranges
* A 12-lead electrocardiogram (ECG) at Screening that is normal or with abnormalities that are considered not clinically significant by the investigator
* Female subjects of childbearing potential must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 prior to first dose of study drug
* Male and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception

Exclusion Criteria:

* HbA1c > 10% at Screening
* Weight loss > 5% weight during the 90 days prior to Screening
* Pregnant or lactating subjects.
* Current alcohol abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* Current substance abuse that is judged by the investigator to potentially interfere with the subject's compliance or safety
* A positive test result for human immunodeficiency virus (HIV-1) antibody, hepatitis B (HBV) surface antigen, or hepatitis C (HCV) antibody
* Unstable cardiovascular disease as defined by any of the following: unstable angina within 6 months prior to Screening; myocardial infarction, coronary artery bypass graft surgery, or coronary angioplasty within 6 months prior to Screening; transient ischemic attack or cerebrovascular accident within 6 months prior to Screening; obstructive valvular heart disease or hypertrophic cardiomyopathy; congestive heart failure (NYHA Class ≥ 2); implanted defibrillator or pacemaker
* Medical history of liver disease, including but not limited to, alcoholic liver disease, autoimmune disorders (e.g., primary biliary cholangitis, primary sclerosing cholangitis, autoimmune hepatitis), drug-induced hepatotoxicity, Wilson disease, clinically significant iron overload, or alpha-1-antitrypsin deficiency. A history of nonalcoholic fatty liver disease (NAFLD), including hepatic steatosis or nonalcoholic steatohepatitis (NASH) is permitted.
* History of intestinal resection or malabsorptive condition that may limit the absorption of study drug
* Presence of severe peptic ulcer, gastroesophageal reflux disease, or other gastric acid hypersecretory conditions at Screening, in the opinion of the investigator
* Any scheduled surgery during the trial period, excluding minor surgical procedures performed under local anesthesia, in the opinion of the investigator
* History of malignancy within 5 years prior to Screening except adequately treated carcinoma in situ of the cervix, and/or squamous cell cancer, or other localized non-melanoma skin cancer
* History of significant drug allergy, such as anaphylaxis or significant drug sensitivity, in the opinion of the investigator
* Known hypersensitivity to study drug, its metabolites, or formulation excipients
* Presence of any medical condition that could, in the opinion of the investigator, compromise the subject's ability to participate in the study, including a history of substance abuse or a psychiatric disorder, including any subject with a psychiatric hospital admission or emergency room visit in the 2 years prior to Screening
* Any laboratory abnormality that in the opinion of the investigator could adversely affect the safety of the subject or impair assessment of study results
* Subjects on any oral medication with a narrow therapeutic window (e.g., warfarin, digoxin, tricyclic antidepressants, lithium, aminophylline, theophylline, and anticonvulsants)
* Medications or therapies prescribed or taken over-the-counter for weight loss, in the 90 days prior to Screening.
* Receipt of vaccination for COVID-19 or any other live vaccine within 14 days of planned dosing of study drug

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in insulin sensitivity | Through study completion, up to Day 84 of the study
  Oral glucose tolerance test will be used to measure insulin sensitivity.
Incidence of TLC-3595 treatment-emergent adverse events | Through study completion, up to Day 84 of the study
  Adverse events (AEs) - severity of the AEs will be graded using the Common Terminology Criteria for AE (CTCAE) (v5.0). The relationship between AEs and the study drug will be indicated as related or not related.

CONTACTS AND LOCATIONS:
Overall Officials: OrsoBio Study Director, Study Director — OrsoBio, Inc
Locations (3):
- New Zealand (3):
  - OrsoBio Research Site, Auckland
  - OrsoBio Reseach Site, Auckland
  - OrsoBio Research Site, Christchurch